CLINICAL TRIAL: NCT02948946
Title: The Clinical Utility of a Blood-Based Multitranscriptome Assay as a Biomarker for Gastroenteropancreatic and Lung Neuroendocrine Tumors
Brief Title: Clinical Utility Assay as a Biomarker for Gastroenteropancreatic and Lung Neuroendocrine Tumors
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-18756
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumor; Lung Neuroendocrine Neoplasm
Keywords: lung cancer; pancreatic cancer
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor; Lung Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neuroendocrine Tumor (NET) Cohort: Participants with histologically or cytologically proven diagnosis of any grade, any stage NET of gastroenteropancreatic (GEP) or lung origin; In the first stage of the study (initial 50 patients) only potential participants with stage IV, well-differentiated tumors (G1/G2) will be enrolled.
  Interventions: Procedure: NETest
- Non-NET Cohort: Participants with histologically or cytologically proven diagnosis of any grade, any stage gastrointestinal (GI) malignancies.
  Interventions: Procedure: NETest

INTERVENTIONS:
Procedure: NETest — 5 mL of blood will be drawn from participants for testing.

SUMMARY:
The purpose of this study is to evaluate how well an investigational blood test performs. The study will look at the sensitivity and specificity of a blood-based multitranscriptome assay (NETest).

ELIGIBILITY:
Inclusion Criteria:

NET Cohort-

* Patients with histologically or cytologically proven diagnosis of any grade, any stage NET of GEP or lung origin; In the first stage of the study (initial 50 patients) only patients with stage IV, well-differentiated tumors (G1/G2) will be enrolled.
* Patients with stable or progressive disease, as documented on a scan (CT, MRI); Progression status will be documented on case report form (CRF).
* Allowed prior therapies include: a.) Surgery (tumor surgery at least four weeks prior to study entry); b.) Locoregional therapy such as: chemoembolization, radio-embolization, radiofrequency ablation, radiotherapy at least six weeks prior to study entry; c.) Any number of previous lines of systemic therapy, providing that cytotoxic therapies (chemotherapy, PRRT) have been discontinued at least 4 weeks prior to study entry.

Non-NET Cohort -

* Healthy participants
* Patients with histologically or cytologically proven diagnosis of any grade, any stage GI malignancies.

Exclusion Criteria:

NET Cohort -

* Patients on treatment with cytotoxic agents (chemotherapy, PRRT).
* Patients with renal insufficiency or congestive heart failure.
* No other active malignancy within 3 years of enrolment except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission.

Non-NET Cohort

* Patients with GI malignancies with neuroendocrine differentiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants to be enrolled in the study will be recruited within the Gastrointestinal (GI) Clinic of Moffitt Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Rate of Successful Test Results Per Cohort | 12 months
  Investigators have designed the study to test the null hypothesis that the NETest has a sensitivity and specificity of 70% or less in NET patients. The sample size calculation has been based on the assumption that a sensitivity and specificity of greater than 90% would generate further interest in the test for unselected NET patients. Power and type 1 error will be 99% and 5% respectively. Under this model, 80 or more positive tests in the cohort of 100 patients with NETs would lead to the rejection of the null hypothesis, suggesting that the NETest is sensitive. Likewise, 80 or more negative tests in 100 patients without NETs will suggest that NETest is specific. An interim analysis will be performed to rule out the futility of the NETest. Futility will be defined as a rate of false positive or false negative >25%. Hence, if 12 or more false positives or negatives are observed among the first 50 participants, the study will be suspended, pending review by the investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Strosberg, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/